CLINICAL TRIAL: NCT01201278
Title: A Phase 1, Randomized, 3-Way Crossover, Investigator Initiated Proof-of-Concept Study to Investigate Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Two Doses of Intranasally Administered Regular Human Insulin Compared to a Single Dose of a Subcutaneously Injected Rapid Acting Insulin Analog (Humalog®) in Subjects With Type I Diabetes
Brief Title: PK/PD Study of Intranasal Insulin in Type I Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hompesch, Marcus, M.D. (Individual)
Collaborators: Profil Institute for Clinical Research, Inc. (Other)
Responsible Party: Hompesch, Marcus, M.D., Profil Institute for Clinical Research, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NI2010-001
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes
Keywords: intranasal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nasal insulin 8 IU (Experimental): Nasal insulin at a dose estimated to be equivalent to 8 IU bioavailable insulin
  Interventions: Drug: Insulin
- Nasal insulin 16 IU (Experimental): Nasal insulin at a dose estimated to be equivalent to 16 IU bioavailable insulin
  Interventions: Drug: Insulin
- Subcutaneous insulin lispro 8 U (Active Comparator): Subcutaneous insulin lispro (Humalog®) 8 U
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: Insulin — Nasal insulin at a dose estimated to be equivalent to 8 IU bioavailable insulin
  Arms: Nasal insulin 8 IU
Drug: Insulin — Nasal insulin at a dose estimated to be equivalent to 16 IU bioavailable insulin
  Arms: Nasal insulin 16 IU
Drug: Insulin LISPRO — Subcutaneous insulin lispro 8 U
  Arms: Subcutaneous insulin lispro 8 U

SUMMARY:
This study is designed to compare the safety and tolerability of two different doses of intranasally administered regular human insulin with those of a single dose of the rapid-acting insulin analog lispro Humalog® after subcutaneous injection. In addition to safety and tolerability, various pharmacokinetic (PK) and pharmacodynamic (PD) parameters will be evaluated by means of the euglycemic glucose clamp technique.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with type 1 diabetes between the ages of 18 and 65 years, inclusive.
2. Type 1 diabetes clinically diagnosed ≥ 12 months.
3. Treated with multiple daily insulin injections ≥ 12 months or an insulin pump.
4. HbA1c ≤ 10 % by local laboratory analysis (one retest within a week is permitted with the result of the last test being conclusive).
5. Fasting serum C-peptide ≤ 0.3 nmol/L.
6. BMI between 18-28 kg/m², inclusive.
7. Signed, written IRB-approved informed consent.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, oncologic, or neurologic (to include history of seizures) disease; hypoglycemic episodes; intercurrent illness (such as influenza); or allergic disease (including severe drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Clinical significance to be determined by the PI.
2. History of recent nose bleed, history of nasal polyps, nasal surgery other than cosmetic rhinoplasty or cauterization.
3. As judged by the investigator, clinically significant findings in laboratory data. (Anemia with hematocrit less than 33% at screening is specifically exclusionary.)
4. Clinically significant abnormal ECG at screening, as judged by the Investigator.
5. Clinically significant abnormalities in vital signs at screening, as judged by the Investigator.
6. Known allergy to trial product or any other ingredient in the study drug.
7. Positive HIV 1 (human immunodeficiency virus) antibody test, hepatitis B (anti-HBsAg) or hepatitis C (anti-HCV) antibody test.
8. History or evidence of alcohol or drug abuse within the past 3 years.
9. History of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in 1st degree relatives (parents, siblings or children) as judged by the Investigator.
10. Use of drugs that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action or glucose utilization.
11. Blood donation or high volume phlebotomy, e.g., >500 mL, within 56 days before dosing.
12. Participation in a study of any investigational drug or device 30 days before enrollment in this study.
13. The subject is unfit for the study in the opinion of the investigator.
14. Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures include sterilization, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomized partner).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Insulin tolerability, PK, and PD | 120 minutes
  To assess safety and tolerability, and to compare the insulin AUC over 0-120 min for each of the three insulin applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States